CLINICAL TRIAL: NCT00940342
Title: Rituximab In Combination With Sargramostim (GM-CSF) In Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Rituximab Plus Sargramostim (GM-CSF) In Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0102; NCI-2012-01670 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-02

CONDITIONS: Leukemia
Keywords: Chronic Lymphocytic Leukemia; Rituximab; Leukemia; Sargramostim; GM-CSF
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treated and Relapsed - Group 1 (Experimental): Participants receive one (1) course of therapy. One course of therapy consists of four (4) doses of Rituximab 375 mg/m2, administered once weekly by vein for 4 weeks along with GM-CSF 250 mcg subcutaneously three times weekly for 8 weeks.
  Interventions: Drug: GM-CSF (Sargramostim); Drug: Rituximab
- Treated and High-Risk for Progression - Group 2 (Experimental): Participants receive one (1) course of therapy. One course of therapy consists of four (4) doses of Rituximab 375 mg/m2, administered once weekly by vein for 4 weeks along with GM-CSF 250 mcg subcutaneously three times weekly for 8 weeks.
  Interventions: Drug: GM-CSF (Sargramostim); Drug: Rituximab
- 70 Years of Age and Refused Chemo - Group 3 (Experimental): Participants receive one (1) course of therapy. One course of therapy consists of four (4) doses of Rituximab 375 mg/m2, administered once weekly by vein for 4 weeks along with GM-CSF 250 mcg subcutaneously three times weekly for 8 weeks.
  Interventions: Drug: GM-CSF (Sargramostim); Drug: Rituximab

INTERVENTIONS:
Drug: GM-CSF (Sargramostim) — 250 mcg injection under the skin, three times a week for eight weeks.
  Other Names: Sargramostim; Leukine
Drug: Rituximab — 375 mg/m^2 administered intravenously once weekly for four weeks
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to learn if giving granulocyte-macrophage colony-stimulating factor (GM-CSF) together with rituximab can improve the ability of rituximab to shrink or slow the growth of Chronic Lymphocytic Leukemia (CLL). The safety of this combination treatment will also be studied.

DETAILED DESCRIPTION:
GM-CSF is a drug designed to stimulate the immune system. It will increase the number of a certain type of blood cell called neutrophils and macrophages.

Rituximab is a drug designed to bind to a protein, called cluster of differentiation antigen 20 (CD20), that is on the surface of the leukemia cells, allowing the leukemia cells to be destroyed by the immune system.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam, including routine blood tests (about 2 tablespoons). A bone marrow aspirate will be collected. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Imaging studies (such as a chest x-ray or CT scans) may be performed. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will receive GM-CSF as an injection under the skin, three times a week for eight weeks. You will receive rituximab by vein, once a week for four weeks. Usually, the first dose of rituximab requires several hours to complete. Later doses should usually be shorter, but may vary according to individual tolerance. Acetaminophen (Tylenol), diphenhydramine hydrochloride (Benadryl), and steroids (hydrocortisone or similar) will be given before rituximab to decrease the risk of side effects. If side effects do occur during the infusion, you will need to stay at the hospital and be observed until the side effects have gone away. Other than that, treatment will be given on an outpatient basis.

During treatment you will have routine blood tests (about 1 tablespoon) once a week. The treatment will take about 8 weeks to be completed. You will be taken off study if your disease gets worse or if the side effects become too severe.

After treatment is over, you will have a complete physical exam, including routine blood tests (about 2 tablespoons). A bone marrow sample will be taken. Imaging studies (such as a chest x-ray or CT scans) may be repeated to evaluate the effect of the treatment. If this treatment has worked for you, your doctor may advise you to receive it again for a second time.

You will then return for post-treatment evaluation every 6 months for 1 year and then once a year for 3 years or until you start a new treatment.

This is an investigational study. GM-CSF and rituximab have been approved by the FDA for clinical use. Their use together in this study, however, is experimental. Up to 130 patients may take part in this study. All patients will be enrolled at M.D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1. Diagnosis of previously treated B-CLL Rai III-IV or earlier stage disease with evidence of "active disease" as defined by the NCI-sponsored working group 1) weight loss of >10% in prior 6 months, 2) extreme fatigue, 3) fever or night sweats without evidence of infection, 4) worsening anemia or thrombocytopenia, 5) progressive lymphocytosis with a rapid lymphocyte doubling time, 6) marked hypogammaglobulinemia or paraproteinemia, 7) lymphadenopathy >5 cm in diameter.
2. Group 2. Diagnosis of previously untreated B-CLL with Rai stage 0-II disease but high risk for progression based on B2-microglobulin >3.0 mg/mL, or with symptoms or significant fatigue.
3. Group 3. Patients age 70 years of age and older with previously untreated B-CLL and Rai stage III-IV or earlier stage disease with indication for treatment who refused chemotherapy.
4. Age 15 years or above.
5. Adequate renal and hepatic functions (creatinine <2.5 mg/dL, bilirubin <2 mg/dL). Patients with renal or liver dysfunction due to organ infiltration by lymphocytes are eligible, as are patients with elevated bilirubin and history consistent with Gilbert's disease.
6. Performance status <3 (Zubrod Scale).
7. No active viral hepatitis

Exclusion Criteria:

1) None.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-10-12 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2004 through January 2007. Of the 130 participants recruited, 119 participants were recruited at The University of Texas (UT) MD Anderson Cancer Center, 6 at The University of California San Diego, and 5 participants were recruited at Dana Farber Cancer Institute.
Groups:
- Untreated and High-Risk for Progression - Group 2; 70 Years of Age and Refused Chemo - Group 3: Participants receive one (1) course of therapy. One course of therapy consists of four (4) doses of Rituximab 375 mg/m2, administered once weekly by vein for 4 weeks along with GM-CSF 250 mcg subcutaneously three times weekly for 8 weeks.
  GM-CSF (Sargramostim): 250 mcg injection under the skin, three times a week for eight weeks.
  Rituximab: 375 mg/m^2 administered intravenously once weekly for four weeks
Period: Overall Study
Arm/Group | Treated and Relapsed - Group 1 | Untreated and High-Risk for Progression - Group 2 | 70 Years of Age and Refused Chemo - Group 3
Started | 50 | 40 | 40
Completed | 50 | 38 | 39
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treated and Relapsed - Group 1 | Untreated and High-Risk for Progression - Group 2 | 70 Years of Age and Refused Chemo - Group 3 | Total
Number analyzed (Participants) | 50 | 40 | 40 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 36 | 0 | 56
  >=65 years | 30 | 4 | 40 | 74
Age, Continuous [Median (Full Range); unit: years] | 68 [41 to 84] | 56.5 [34 to 70] | 73 [70 to 83] | 69 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 14 | 49
  Male | 34 | 21 | 26 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 7
  White | 49 | 38 | 36 | 123
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 40 | 40 | 130

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate - Complete Response (CR) + Partial Response (PR). CR is the absence of Lymphocyte infiltrates on biopsy, <30% Lymphocytes on Bone Marrow Aspirate, Lymphocytes < 4,000ul , Hemoglobin >11.0 g/dl , Platelets >1000,000/ul, Polymorphonuclear neutrophils (PMN) >1,500/ul, Liver/Spleen not palpable, Nodes none. PR is <30% Lymphocytes with residual disease on biopsy for nodular PR, Lymphocytes >50% decrease, Hemoglobin (un-transfused) > 11.0 g/dl or >50% improvement from baseline, Platelets > 100,000/ul or 50% improvement from baseline, PMN >1,500 ul or 50% improvement from baseline, Liver/Spleen >/= 50% decrease, Nodes >/= 50%.
Time Frame: Blood tests once a week during 8 weeks of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated and Relapsed - Group 1 | Untreated and High-Risk for Progression - Group 2 | 70 Years of Age and Refused Chemo - Group 3
Number analyzed (Participants) | 50 | 38 | 39
Participants | 23 | 31 | 23

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent and will be followed to resolution or stabilization. Adverse events reported during each treatment course, up to 8 weeks
Arm/Group | Treated and Relapsed - Group 1 | Untreated and High-Risk for Progression - Group 2 | 70 Years of Age and Refused Chemo - Group 3
All-Cause Mortality (participants affected / at risk) | 3/50 | 0/40 | 1/40
Serious Adverse Events (participants affected / at risk) | 5/50 | 3/40 | 4/40
Other Adverse Events (participants affected / at risk) | 21/50 | 16/40 | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated and Relapsed - Group 1 (N=50) | Untreated and High-Risk for Progression - Group 2 (N=40) | 70 Years of Age and Refused Chemo - Group 3 (N=40)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenic Fever (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated and Relapsed - Group 1 (N=50) | Untreated and High-Risk for Progression - Group 2 (N=40) | 70 Years of Age and Refused Chemo - Group 3 (N=40)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10) | 10 (10)
Pain (General disorders) | 4 (4) | 4 (4) | 1 (1)
Fever (General disorders) | 3 (3) | 1 (1) | 1 (1)
Chills (General disorders) | 3 (3) | 0 (0) | 1 (1)
Neutropenia (Infections and infestations) | 11 (11) | 4 (4) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 2 (2)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No